CLINICAL TRIAL: NCT02989883
Title: Clinical Outcomes of Peroral Endoscopic Myotomy for Esophageal Outflow Obstruction
Brief Title: Clinical Outcomes of Peroral Endoscopic Myotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hwoon-Yong Jung, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0999
Record Dates: First submitted 2016-12-04; First posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Achalasia
Keywords: achalasia; POEM; outcome
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peroral endoscopic myotomy (POEM) (Other): Patients who received POEM
  Interventions: Other: peroral endoscopic myotomy

INTERVENTIONS:
Other: peroral endoscopic myotomy — The procedure consists of four steps: 1) mucosal incision 10-15 cm above the esophagogastric junction to allow entry into the submucosa, 2) creation of a submucosal tunnel until the lower esophageal sphincter is reached, 3) myotomy of the circular muscle layer, and 4) closure of the mucosal entry with endoclips.

SUMMARY:
Esophageal outflow obstruction is characterized by failure to relax the lower esophageal sphincter (LES), resulting in impaired flow of ingested food into the stomach. The subsequent stasis of ingested food leads to symptoms of dysphagia, regurgitation, chest pain, and weight loss. The core objective of the treatment of esophageal outflow obstruction is to disrupt the LES and reduce its pressure to allow esophageal emptying. Therapeutic options include pharmacologic therapy, Botulinum toxin injection, pneumatic balloon dilation, and surgical myotomy with partial fundoplication. In addition, peroral endoscopy myotomy (POEM) has recently been introduced as a minimally invasive treatment, but there have a few studies regarding long-term outcomes. The aim of this study is to evaluate clinical outcomes of POEM for esophageal outflow obstruction.

DETAILED DESCRIPTION:
Prospective study

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed as esophageal outflow obstruction
* Patients with informed consent

Exclusion Criteria:

* Diagnostic uncertainty
* Patients who are not suitable for general anesthesia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-03 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
number of patients with Eckardt score <3 after the procedure | 1 month after the procedure

SECONDARY OUTCOMES:
adverse events which are related to the procedure | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Hwoon-Yong Jung, Principal Investigator — Asan Medical Center
Locations (1):
- Department of Gastroenterology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gong EJ, Na HK, Ahn JY, Jung KW, Kim DH, Choi KD, Song HJ, Jung HY. Prospective evaluation of the efficacy of peroral endoscopic myotomy in patients with achalasia. Medicine (Baltimore). 2021 Jun 11;100(23):e26248. doi: 10.1097/MD.0000000000026248. PMID 34115014